CLINICAL TRIAL: NCT03993041
Title: Telehealth Psychotherapy for Depression in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Alice Cronin-Golomb, Director, Vision & Cognition Laboratory, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5222
Record Dates: First submitted 2019-06-16; First posted 2019-06-20 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Depression; Parkinson's Disease
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioral therapy (CBT) (Experimental): Individuals in the CBT arm are expected to participate in a phone screen + baseline phase (one assessment) + 10-12 weeks of CBT intervention + post-intervention assessment + 6 week follow-up assessment.
  Interventions: Behavioral: Cognitive-behavioral therapy (CBT)
- Waitlist Control (Active Comparator): Individuals in the Waitlist Control arm are expected to participate in a phone screen + baseline phase (two assessments, 12 weeks apart) + 10-12 weeks of CBT intervention + post-intervention assessment + 6 week follow-up assessment.
  Interventions: Behavioral: Cognitive-behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy (CBT) — Study therapists will deliver cognitive-behavioral therapy (CBT) based on an emotion-focused, transdiagnostic protocol. CBT targets problematic thoughts, feelings, and behaviors through goal-oriented, systematic procedures. The intervention used in this study is designed to target emotional processing with an emphasis on present-focused awareness, cognitive flexibility, emotional avoidance, awareness and tolerance of physical sensations, and situation-based emotion exposure. The intervention is designed to help individuals better understand emotional experiences in order to respond to intense emotions in a more adaptive way.

SUMMARY:
Depression is a prevalent non-motor symptom of Parkinson's disease (PD). Cognitive-behavioral therapy (CBT) has been shown to be an effective treatment for depression in PD. CBT is usually administered in-person in weekly sessions, but PD motor disability, stigma, and transportation issues may prevent attending such therapy sessions. CBT administered via live videoconference technology may allow the treatment of depression, while circumventing the barriers that deter those with PD from seeking psychological services. The investigators propose that videoconference CBT will improve mood in individuals with PD who have depression.

DETAILED DESCRIPTION:
The investigators plan to conduct a randomized control trial with 12 participants. Six (PD-early) will receive three assessments: baseline, immediately post-treatment (post1), and 6 weeks after treatment (post2). The other six (PD-waitlist) will have an additional assessment (Baseline 2; 12 weeks after Baseline 1) to examine practice effects before beginning treatment, and then will have the post1 and post2 assessments (four assessments).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (PD), any subtype
* Depression
* Internet access and a webcam
* For psychotropic and dopaminergic medications, participants may enroll only if they are stable for at least 6 weeks and 2 weeks, respectively, before beginning the study
* The investigators will enroll only depressed individuals with PD who are not already receiving or are willing to stop other ongoing psychotherapy before beginning this treatment study

Exclusion Criteria:

* Serious chronic medical or neurological illness, other than PD
* History of traumatic brain injury
* Mental retardation
* Current or recent (past 90 days) history of substance abuse or drug dependence, with the exception of nicotine, marijuana, and caffeine
* Active suicidal or homicidal ideation or intent
* Dementia
* Current DSM-5 diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or substance/medication-induced disorder
* Previous experience with an adequate trial of cognitive-behavioral therapy (8 sessions within the past 5 years
* Concurrent psychosocial treatment (i.e., therapy) focused on depression, anxiety, or other related disorders, or are not willing to refrain from initiating additional therapy during the study
* Concurrent psychotropic medications if not stabilized or not willing to maintain a stable dosage of psychotropic medications, such as medications for depression or anxiety, during study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Anxiety and Related Disorders Interview Schedule for DSM-5 | Change in diagnosis of depression from baseline to post-treatment (approximately 12 weeks after baseline) and 6-week follow-up.
  Semi-structured diagnostic interview for assessment of mood and related disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cronin-Golomb, Ph.D., Principal Investigator — Boston University
Locations (1):
- Vision & Cognition Laboratory, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No